CLINICAL TRIAL: NCT01333228
Title: Pilot Clinical Trial (Phase I/II) to Evaluate Safety and Therapeutic Effects of the Administration of Autologous Bone Marrow-derived EPCs in Patients With Advanced Liver Cirrhosis
Brief Title: Evaluate Safety and Efficacy of Autologous Bone Marrow-derived Endothelial Progenitor Cells in Advanced Liver Cirrhosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Foundation Ramon Areces (Unknown); Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPC/CIRR
Record Dates: First submitted 2011-04-01; First posted 2011-04-11 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endothelial Progenitors Cells (Experimental): Autologous bone marrow-derived endothelial progenitor cells
  Interventions: Other: Autologous bone marrow-derived endothelial progenitor cells

INTERVENTIONS:
Other: Autologous bone marrow-derived endothelial progenitor cells — Intraarterial administration (hepatic artery) of autologous bone marrow-derived endothelial progenitor cells

SUMMARY:
Endothelial Progenitor Cells (EPC) represent a small cellular population of bone marrow and peripheral blood cells. EPCs are recruited into injured tissues and play an important role in regeneration and reparation. Experimental and clinical data suggest that EPCs have hepatoprotective activity and could improve liver regeneration during acute and chronic liver injury. The aim of this project is to evaluate the safety and therapeutic effects of autologous bone marrow-derived EPCs, when administered through the hepatic artery of patients with advanced liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis (Child-Pugh 8 or above).
* Ability to sign informed consent

Exclusion Criteria:

* Age <18 or >75
* Variceal bleeding or severe infection within the past 30 days before screening
* Chronic encephalopathy preventing the ability to sign informed consent (it could be done by legal representant of the patient) and/or the ability to follow the study protocol
* Hepatocellular carcinoma (previous or current)
* Any current or previous malignancy (within 5 years before the inclusion) except "in situ" tumors or skin basal cell carcinomas
* Any severe extrahepatic disease during the past 30 days before the inclusion
* Any current decompensated chronic disease
* Any contraindication for the examinations of the clinical protocol (medullar aspiration, arteriography, HVPG measurement)
* Any other condition that could negatively affect the compliance with the protocol
* Pregnant or breast-feeding women
* Participation in a trial of an experimental drug or device within 30 days before screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-06; Primary Completion 2014-10 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and tolerability | 12 months
  The safety of the administration of autologous bone marrow-derived EPC in patients with advanced cirrhosis will be evaluated by anamnesis, physical examination, hematological and biochemical variables and imaging examination.

SECONDARY OUTCOMES:
Changes of liver function test as a measure of the effect on liver function | 12 months
  Determination of liver function test (aminotransferases,albumin, bilirubin and protrombin time) and calculation of Model for End-Stage Liver Disease (MELD) and Chil-Pugh scores. Differences in these variables compared to baseline will be considered as a measure of the effect on liver function.
Effect on portal hypertension | 12 months
  Changes in Hepatic Venous Pressure Gradient (HVPG) will be used to assess the effect on portal hypertension.
Effect on complications of liver cirrhosis | 12 months
  Ascitis grade, episodes of upper gastrointestinal bleeding as well as of episodes of hepatic encephalopathy will be used as a measure of the effect of the treatment on the complications of liver cirrhosis.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Quiroga, MD, PhD, Principal Investigator — Liver Unit, Clinica Universidad de Navarra/Centro de Investigación Biomédica en Red en el Área temática de Enfermedades Hepáticas y Digestivas (CIBERehd)(Pamplona-Spain); Jesus Prieto, MD, PhD, Study Chair — Liver Unit, Clinica Universidad de Navarra/Centro de Investigación Biomédica en Red en el Área temática de Enfermedades Hepáticas y Digestivas (CIBERehd)/Centro de Investigación Medica Aplicada (CIMA)(Pamplona-Spain); Delia D'Avola, MD, Study Chair — Liver Unit, Clinica Universidad de Navarra/Centro de Investigación Biomédica en Red en el Área temática de Enfermedades Hepáticas y Digestivas (CIBERehd)(Pamplona-Spain); Jose Ignacio Herrero, MD, PhD, Study Chair — Liver Unit, Clinica Universidad de Navarra/Centro de Investigación Biomédica en Red en el Área temática de Enfermedades Hepáticas y Digestivas (CIBERehd)(Pamplona-Spain); Bruno Sangro, MD, PhD, Study Chair — Liver Unit, Clinica Universidad de Navarra/Centro de Investigación Biomédica en Red en el Área temática de Enfermedades Hepáticas y Digestivas (CIBERehd)(Pamplona-Spain); Veronica Fernandez Ruiz, PhD, Study Chair — Centro de Investigación Medica Aplicada (CIMA)(Pamplona-Spain); Javier Perez Calvo, MD,PhD, Study Chair — Hematology, Clinica Universidad de Navarra (Pamplona-Spain); Mercedes Iñarrairaegui, MD PhD, Study Chair — Liver Unit, Clinica Universidad de Navarra/Centro de Investigación Biomédica en Red en el Área temática de Enfermedades Hepáticas y Digestivas (CIBERehd)(Pamplona-Spain); Jose Ignacio Bilbao, MD,PhD, Study Chair — Radiology, Clinica Universidad de Navarra (Pamplona-Spain)
Locations (1):
- Clinica Universidad de Navarra, Pamplona, Navarre, Spain

REFERENCES:
- [Derived] D'Avola D, Fernandez-Ruiz V, Carmona-Torre F, Mendez M, Perez-Calvo J, Prosper F, Andreu E, Herrero JI, Inarrairaegui M, Fuertes C, Bilbao JI, Sangro B, Prieto J, Quiroga J. Phase 1-2 pilot clinical trial in patients with decompensated liver cirrhosis treated with bone marrow-derived endothelial progenitor cells. Transl Res. 2017 Oct;188:80-91.e2. doi: 10.1016/j.trsl.2016.02.009. Epub 2016 Feb 24. PMID 26972567
- See also: Clinica Universidad de Navarra — http://www.cun.es
- See also: Centro de Investigación Biomédica en Red en el Área temática de Enfermedades Hepáticas y Digestivas — http://www.ciberehd.org